CLINICAL TRIAL: NCT00805597
Title: A Phase Ⅲ Randomized Clinical Trial of Postmastectomy Radiotherapy in Breast Cancer With One to Three Positive Nodes
Brief Title: Clinical Trial of Postmastectomy Radiotherapy in Breast Cancer With One to Three Positive Nodes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The recuiting was to slow to complete the study
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shu lian Wang, M.D., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2008B06
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; mastectomy; one to three positive nodes; radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy (Experimental): radiotherapy of 50Gy/25/f/5w to the ipsilateral chest wall and supraclavicular region
  Interventions: Radiation: radiation
- no radiotherapy (Active Comparator): no radiotherapy
  Interventions: Radiation: no radiation

INTERVENTIONS:
Radiation: radiation — radiotherapy of 50Gy/25f/5w to the chest wall and supraclavicular nodal region
  Arms: radiotherapy
Radiation: no radiation — no radiotherapy
  Arms: no radiotherapy

SUMMARY:
The purpose of this study is to evaluate postmastectomy radiotherapy in breast cancer patients with one to three positive nodes.

DETAILED DESCRIPTION:
Eligible breast cancer patients with mastectomy and axillary dissection are randomized into 2 groups:radiotherapy of 50 Gy in 25 fractions within 5 weeks to ipsilateral chest wall and supraclavicular nodal region,and no radiotherapy.

During and after radiotherapy, the patients are followed and the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Ipsilateral histologically confirmed invasive breast cancer
* Undergone total mastectomy and axillary dissection
* T1-2 and one to three axillary lymph nodes positive
* A minimum of 10 axillary nodes dissected
* Fit for chemotherapy(if indicated),endocrine therapy(if indicated)and postoperative irradiation
* Written,informed consent

Exclusion Criteria:

* Patients who undergone previous irradiation to the ipsilateral chest wall and supraclavicular region
* Previous or concurrent malignant other than non-melanomatous skin cancer
* Unable or unwilling to give informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
overall survival | 10 years

SECONDARY OUTCOMES:
loco-regional recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye-xiong Li, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China